CLINICAL TRIAL: NCT05196139
Title: Visual Outcome After Vitrectomy With Subretinal tPA Injection to Treat Submacular Hemorrhage Secondary to Age-related Macular Degeneration or Macroaneurysm
Brief Title: Visual Outcome After Vitrectomy With Subretinal tPA Injection
Acronym: EVA-tPA
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 65203
Record Dates: First submitted 2021-12-24; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective study — vitrectomy performed in case of submacular bleeding

SUMMARY:
evaluate the safety of Eva surgical system

DETAILED DESCRIPTION:
The purpose of this retrospective study is to evaluate the safety and clinical results using this surgical technique when performed using the EVA surgical system and associated instrumentation and disposable surgical equipment

ELIGIBILITY:
Inclusion Criteria:

* patients with VTX subretinal tPA ( + phaco)
* patients with submacular bleeding

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgery on the patients included in the study will have been performed using the EVA surgical system (DORC).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
pre-operative best corrected visual acuity | pre surgery
  • The pre-operative BCVA will be taken from the visit when the indication for the surgery was set
Surgical adverse events | postoperative visit on day 1
  Surgical adverse events or issues that were recorded in the surgical report
post-operative best corrected visual acuity | 6 weeks after surgery
  The post-operative BCVA will be taken from the latest visit after the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No